CLINICAL TRIAL: NCT03972631
Title: Lifestyle Interventions for the Treatment of Non-alcoholic Fatty Liver Disease in Overweight and Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Liu Zhong, Clinical Professor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHPF2018-NALFD-1
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: Lifestyle interventions; Low-carbohydrate diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle education (Placebo Comparator): The participants in this group will be provided usual recommendation, including the diet principles, activity guideline and behavioral strategies at baseline. In addition, the participants will have access to an APP, with which the participants could learn more information of body weight management, and keep records of diet, activity and body weight during the study.
  Interventions: Behavioral: Lifestyle education
- Intensive Lifestyle Intervention (Experimental): The participants in this group will be provided a comprehensive intervention, including goal setting, one to one support by the lifestyle counselors, and meal replacement products, in addition to the information and APP which are provided to the Lifestyle education group.
  Interventions: Behavioral: Lifestyle education; Behavioral: Intensive lifestyle intervention; Behavioral: Hypocaloric low-carbohydrate diet plan

INTERVENTIONS:
Behavioral: Lifestyle education — Lifestyle education include the diet principles, physical activity guideline and behavioral strategies.
Behavioral: Intensive lifestyle intervention — One to one intensive lifestyle intervention according to the diet and activity plan
  Arms: Intensive Lifestyle Intervention
Behavioral: Hypocaloric low-carbohydrate diet plan — A diet plan with restricted calorie and carbohydrate intake
  Arms: Intensive Lifestyle Intervention

SUMMARY:
Lifestyle intervention is the most important management of non-alcoholic fatty liver diseases (NAFLD) patients. Weight reductions of 5-10% can improve non-alcoholic steatosis and fibrosis. However, the options for treatment in the clinics are limited. Therefore, in this study, we investigated the effectiveness of different lifestyle intervention strategies in NAFLD patients.

DETAILED DESCRIPTION:
This is a multicenter, randomized clinical trial nested within a cohort study in overweight and obese non-alcoholic fatty liver diseases (NAFLD) patients. In this study, 1500 eligible patients will be recruited, and demographic information and clinical data will be collected at baseline. Among these, 292 participants who agree to be randomized will be randomized into two intervention groups, including lifestyle education (LE), and intensive lifestyle intervention with low-carbohydrate diet (ILI), aiming to induce a loss ≥ 10% of initial weight in 3 months. The remainder will chose the treatment which they prefer according to the clinical practice. At the 3th, 6th and 12th month, all the participants will be followed, and data will be collected to study the development of NAFLD in different lifestyle intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Man or women aged 18-65 years;
* Confirmed diagnosis of NAFLD according to the 2018 Chinese Guidelines for Prevention and Treatment of NAFLD;
* Body mass index (BMI)of 25.0 to 35.0 kg/m2;
* Patients without medicine for treatment of NAFLD;

Exclusion Criteria:

* Patients with other diseases that can lead to fatty liver;
* Patients use amiodaron, methotrexate, tamoxifen, glucocorticoid, estrogen, and the other medications that affect weight within 3 months;
* Patients with serious liver dysfunction (AST or/and ALT >3 times of the upper limit of normal), or renal dysfunction (serum creatinine >the upper limit of normal);
* Patients with diseases that need control of dietary protein intake;
* Patients with diseases that affect food digestion and absorption;
* Patients with diagnosed diabetes or those with significantly elevated blood glucose (fasting blood glucose ≥7.0 mmol/L and/or random blood glucose ≥11.1 mmol/L);
* Patients with severe cardiovascular and cerebrovascular diseases or severe hypertension (Grade 3); anemia; mental illness or memory disorder; epilepsy or antiepileptic treatment;
* Patients with secondary obesity;
* Patients with cancer, active tuberculosis, AIDS and other infectious diseases;
* Pregnancy or lactation;
* Physical disability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in BMI | baseline, 3 month
Change in liver function biomarkers | baseline, 3 month
  ALT, AST
Liver Stiffness Measurement | baseline, 3 month
  LSM is suggested as degree of liver fibrosis
Fast Ultrasound Attenuation Parameter | baseline, 3 month
  FAP is suggested as degree of liver steatosis.

SECONDARY OUTCOMES:
Change in BMI | 6 month, 12 month
Change in liver function biomarkers | 6 month, 12 month
  ALT, AST
Change in blood pressure | baseline, 3 month
Change in lipid | baseline, 3 month
  triglyceride, total cholesterol , LDL-C, and HDL-C
Change in glycemic markers | baseline, 3 month
  fasting glucose, fasting insulin, HbA1C
Change in body composition | baseline, 3 month
  muscle mass, fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Zhong, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Z, Jin P, Liu Y, Zhang Z, Wu X, Weng M, Cao S, Wang Y, Zeng C, Yang R, Liu C, Sun P, Tian C, Li N, Zeng Q. A comprehensive approach to lifestyle intervention based on a calorie-restricted diet ameliorates liver fat in overweight/obese patients with NAFLD: a multicenter randomized controlled trial in China. Nutr J. 2024 Jun 13;23(1):64. doi: 10.1186/s12937-024-00968-8. PMID 38872173
- [Derived] Sun P, Huang L, Shuai P, Wan Z, Liu Y, Xue J, Liu Y. Effect of a High Protein, Low Glycemic Index Dietary Intervention on Metabolic Dysfunction-Associated Fatty Liver Disease: A Randomized Controlled Trial. Front Nutr. 2022 Apr 27;9:863834. doi: 10.3389/fnut.2022.863834. eCollection 2022. PMID 35571881